CLINICAL TRIAL: NCT05597358
Title: Efficacy of High Intensity Laser Therapy for Reducing Pain During Intercourse in Women with Provoked Vestibulodynia: a Multicenter Randomized Controlled Trial
Brief Title: Efficacy of High Intensity Laser for Provoked Vestibulodynia
Acronym: Laser_RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Exogenia (Unknown); CHU de Quebec-Universite Laval (Other); Kinatex l'Ormière (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-31-2023-4770
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Vulvodynia
Keywords: Laser; Provoked vestibulodynia; Pain; Sexual dysfunctions
MeSH Terms: conditions — Vulvodynia; Pain | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: * Baseline evaluation
  * Randomization to active laser or sham laser (12 sessions in 6 consecutive weeks) Post-treatment evaluation (2 weeks post-treatment)
  * Follow-up evaluation (6 months post-treatment)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, outcomes assessors and data analysts will be masked to group assignation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Intensity Laser Therapy (HILT) (Active Comparator): Active high intensity laser therapy for 12 biweekly sessions (6 consecutive weeks of biweekly treatments)
  Interventions: Radiation: High Intensity Laser Therapy (HILT)
- Sham High Intensity Laser Therapy (Sham Comparator): Sham high-intensity laser therapy for 12 biweekly sessions (6 consecutive weeks of biweekly treatments)
  Interventions: Radiation: Sham High Intensity Laser Therapy

INTERVENTIONS:
Radiation: High Intensity Laser Therapy (HILT) — Nd:Yag 1064 nm pulsed high intensity laser will be applied to the vulvar area.
  Other Names: Nd:Yag laser
  Arms: High Intensity Laser Therapy (HILT)
Radiation: Sham High Intensity Laser Therapy — Nd:Yag 1064 pulsed high intensity laser deactivated probe will be applied to the vulvar area.
  Other Names: Sham; Control; Deactivated probe
  Arms: Sham High Intensity Laser Therapy

SUMMARY:
This is a multicenter randomized controlled trial (RCT) investigating the effects of laser treatments in women suffering from provoked vestibulodynia compared to a sham-laser treatment. Following their enrollment in the study, participants will undergo a gynecological examination for confirmation of their diagnoses. Eligible participants will then be asked to complete a consent form and the baseline assessment. The baseline assessment consists of the completion of validated questionnaires (outcome measures). Participants will be randomized into the laser group or sham-laser group. The laser group will receive 12 sessions of active high intensity laser therapy (HILT) (30 minutes biweekly for 6 consecutive weeks). The sham-laser group will receive 12 sessions (30 minutes biweekly for 6 consecutive weeks) of laser therapy using a deactivated probe. Outcome measures (validated questionnaires) will also be assessed 2 weeks post-treatment as well as 6 months post-treatment (follow-up assessment).

DETAILED DESCRIPTION:
Vulvodynia, a chronic vulvar pain condition, affects between 8 and 18% of reproductive-aged women. The main subtype of vulvodynia is provoked vestibulodynia (PVD), which is characterized by a sharp or burning pain at the vaginal opening while applying pressure to the vulvar vestibule or attempting vaginal penetration. Women suffering from PVD experience greater psychological distress, a worsened quality of life and overall well-being as well as sexual dysfunctions for both the women and their intimate partners. Women suffering from PVD have limited treatment options, and some women have persistent pain despite the available treatment options. Therefore, a new therapeutic avenue needs to be explored. High intensity laser therapy (HILT), a non-invasive and non-ablative laser technique, was found to be effective in several chronic pain conditions. Our randomized pilot study confirmed that HILT is feasible for treating PVD. The promising findings obtained provided support for conducting this large multicenter randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe pain (≥ 5/10) at least 90% of the time during sexual intercourse or attempted sexual intercourse for at least 3 months
* Provoked vestibulodynia of at least 3 months duration prior to the study and diagnosed by a standardized gynaecologic exam

Exclusion Criteria:

* Other causes of vulvovaginal pain (e.g., spontaneous vulvovaginal pain not related to sexual intercourse/contact, dermatological condition, herpes, vulvovaginal atrophy)
* Post-menopausal state
* Current pregnancy or pregnancy in the last year
* Urogynecological condition (e.g., pelvic organ prolapse (POP) ≥ 3, urinary/vaginal infection active or in the last 3 months)
* Anterior vulvar, vaginal or pelvic surgery (e.g., vestibulectomy, corrective pelvic organ prolapse surgery)
* Prior use of laser treatments for vulvar pain
* Expected changes of medication that could influence pain perception (e.g., analgesic, antidepressant)
* Other medical conditions that could interfere with the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity during intercourse | Baseline, 2-week post-treatment evaluation, 6-months follow-up assessment
  To explore changes in pain intensity during intercourse (Numerical Rating Scale (NRS), ranging from 0 to 10, where 0 is no pain at all, and 10 is the worst pain ever)

SECONDARY OUTCOMES:
Change in pain quality | Baseline, 2-week post-treatment evaluation, 6-months follow-up assessment
  To explore changes in the sensory, affective, and evaluative components of pain (McGill-Melzack Questionnaire). Minimum value: 0, Maximum value: 78, higher scores indicate a worse outcome (higher pain).
Change in sexual function | Baseline, 2-week post-treatment evaluation, 6-months follow-up assessment
  To explore changes in sexual function (Female Sexual Function Index - FSFI). Minimum value: 2, Maximum value: 36, lower scores indicate a worse outcome (low sexual function).
Change in sexual distress | Baseline, 2-week post-treatment evaluation, 6-months follow-up assessment
  To explore changes in sexual distress (Female Sexual Distress Scale - FSDS). Minimum value: 0, Maximum value: 52, higher scores indicate a worse outcome (higher sexually-related distress).
Change in pain catastrophizing | Baseline, 2-week post-treatment evaluation, 6-months follow-up assessment
  To explore changes in pain catastrophizing (Pain Catastrophizing Scale - PCS). Minimum value: 0, Maximum value: 52, higher scores indicate a worse outcome (higher pain catastrophizing).
Change in fear of pain | Baseline, 2-week post-treatment evaluation, 6-months follow-up assessment
  To explore changes in fear of pain (Pain Anxiety Symptoms Scale - PASS-20). Minimum value: 0, Maximum value: 100, higher scores indicate a worse outcome (higher fear of pain).
Change in cognitions regarding vaginal penetration | Baseline, 2-week post-treatment evaluation, 6-months follow-up assessment
  To explore the cognitions of women towards vaginal penetration (Vaginal penetration cognition questionnaire (VPCQ)). Minimum value: 0, Maximum value: 240, higher scores show higher levels of perceived penetration control.
Change in the life impact of pelvic pain | Baseline, 2-week post-treatment evaluation, 6-months follow-up assessment
  To explore the change in the life impact of pelvic pain (Pelvic Pain Impact Questionnaire). Minimum value: 0, Maximum value: 32, higher scores indicate that the pelvic pain of the participants has a strong impact on their life.
Change in intercourse self-efficacy | Baseline, 2-week post-treatment evaluation, 6-months follow-up assessment
  To explore the change self-efficacy regarding painful intercourse (Painful Intercourse Self-Efficacy Scale). Minimum value: 20, Maximum value: 100, higher scores indicate higher self-efficacy.
Level of satisfaction with treatment | 2-week post-treatment evaluation, 6-months follow-up assessment
  To determine acceptability by measuring the participants' satisfaction with the treatment on a Numeric Rating Scale (NRS) ranging from 0 (completely dissatisfied) to 10 (completely satisfied).
Patient's global impression of change | 2-week post-treatment evaluation, 6-months follow-up assessment
  To examine patient self-reported improvement (Patient's Global Impression of Change - PGIC) ranging from "very much worse" to "very much improved" on a 7-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Morin, PT, PhD, Principal Investigator — Université de Sherbrooke
Locations (4):
- Canada (4):
  - Centre Hospitalier Universitaire de Québec - Université Laval, Québec, Quebec
  - Kinatex l'Ormière, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Exogenia, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data will be made available upon approval by the principal investigator and study team.